CLINICAL TRIAL: NCT03257878
Title: Comparative Study Between Systemic Sclerosis and Other Rheumatic Diseases for Health-related Quality of Life in Korean Patients
Brief Title: Health-related Quality of Life in Korean Patients With Rheumatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor, Seoul National University Hospital
Other Study IDs: H-1701-023-821
Record Dates: First submitted 2017-08-11; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-04

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Systemic sclerosis (SSc): validated Korean version of the SF36 and EQ-5D
  Interventions: Other: validated Korean version of the SF36 and EQ-5D
- Rheumatoid arthritis (RA): validated Korean version of the SF36 and EQ-5D
  Interventions: Other: validated Korean version of the SF36 and EQ-5D
- Systemic lupus erythematosus (SLE): validated Korean version of the SF36 and EQ-5D
  Interventions: Other: validated Korean version of the SF36 and EQ-5D
- Sjogren's syndrome: validated Korean version of the SF36 and EQ-5D
  Interventions: Other: validated Korean version of the SF36 and EQ-5D
- Control: validated Korean version of the SF36 and EQ-5D
  Interventions: Other: validated Korean version of the SF36 and EQ-5D

INTERVENTIONS:
Other: validated Korean version of the SF36 and EQ-5D — This is an observational prospective study. SF36 consists of 36 questions that measure patient's HRQoL in 8 domains: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH) that represent the physical HRQoL, vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH) that represent the mental HRQoL. Each domain is scored from 0 (worst health status) to 100 (best health status). The scores of these domains are summarized into the physical component score (PCS) and mental component score (MCS).
  The EQ-5D questionnaire is made up for 2 components; health state description and evaluation. In description part, health status is measured in terms of 5 dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).

SUMMARY:
To compare the health related quality of life of patients with systemic sclerosis with other rheumatic diseases, such as rheumatoid arthritis, systemic lupus erythematosus and Sjogren's syndrome.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a connective tissue disease characterized by vasculopathy, fibrosis, and autoimmunity. The prognosis of the disease depends on the nature and severity of organ involvement. Patients with SSc suffer from digital ulceration, arthritis, progressive skin tightening, and joint contractures that cause pain and limitation of limb function. The cardiopulmonary system may also be severly affected by SSc in the form of interstitial lung disease and pulmonary arterial hypertension, which leads to reduction in exercise capacity and symptomatic dyspnea. Gastrointestinal involvement by SSc may cause malnutrition, and SSc renal crises may result in renal failure. In addition, cosmetic disfigurement resulting from facial and limb skin involvement may lead to social isolation, mood problems, and significant work disability.

It has been reported that health related quality of life (HRQoL) is significantly impared in SSc patients compared to the general population. Moreover, the degree of impairment in SSc patients was comparable to those who suffered from other chronic illnesses such as heart and lung disease, hypertension, diabetes mellitus, and depression. However, there were no studies yet comparing the HRQoL of SSc patients with other rheumatic diseases, such as rheumatoid arthritis (RA) and systemic lupus erythematosus (SLE). Especially, information regarding the impact of SSc on functioning and HRQoL in Korean patients is lacking.

Therefore, the investigators plan to compare the functioning and HRQoL of patients with SSc with other rheumatic diseases, such as RA, SLE, and Sjogrens's syndrome, and healthy controls. A validated Korean version of the Medical Outcomes Study Short Form 36 (SF36) questionnaire and the EuroQol five dimensions questionnaire (EQ-5D) will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 18 years at time of consent
* Patients able to understand written and spoken Korean
* Patients who have been informed about the research
* Patients with SSc meeting the 1980 ACR criteria or 2013 ACR/EULAR criteria for SSc
* Patients with RA meeting the 2010 ACR/EULAR criteria
* Patients with SLE meeting the 1997 ACR criteria or 2012 SLICC criteria
* Patients with Sjogren's syndrome meeting the 2002 AECG criteria or 2012 ACR criteria
* Controls : without any rheumatic diseases

Exclusion Criteria:

* Severe mental retardation
* Any impairment of ability to understand making self-evaluation impossible (using a validated Korean version of the SF36 and EQ-5D)
* Anyone with other rheumatic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Rheumatology clinic at Seoul National University Hospital from March 2017 through to December 2017
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
comparison of physical component scores (PCS) of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion

SECONDARY OUTCOMES:
comparison of mental component scores (MCS) of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of physical functioning (PF) scores of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of physical role (PR) scores of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of bodily pain (BP) scores of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of general health (GH) scores of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of vitality (VT) scores of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of social functioning (SF) scores of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of emotional role (ER) scores of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of mental health (MH) scores of the SF 36 questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion
comparison of the scores of the EQ-5D questionnaire between patients with systemic sclerosis and other rheumatic diseases | once at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Eun Bong Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hudson M, Thombs BD, Steele R, Panopalis P, Newton E, Baron M; Canadian Scleroderma Research Group. Quality of life in patients with systemic sclerosis compared to the general population and patients with other chronic conditions. J Rheumatol. 2009 Apr;36(4):768-72. doi: 10.3899/jrheum.080281. Epub 2009 Feb 17. PMID 19228662
- [Background] Georges C, Chassany O, Toledano C, Mouthon L, Tiev K, Meyer O, Ilie D, Rambeloarisoa J, Marjanovic Z, Cabane J, Sereni D, Pouchot J, Farge D. Impact of pain in health related quality of life of patients with systemic sclerosis. Rheumatology (Oxford). 2006 Oct;45(10):1298-302. doi: 10.1093/rheumatology/kel189. Epub 2006 Jun 4. PMID 16754629
- [Background] Del Rosso A, Boldrini M, D'Agostino D, Placidi GP, Scarpato A, Pignone A, Generini S, Konttinen Y, Zoppi M, Vlak T, Placidi G, Matucci-Cerinic M. Health-related quality of life in systemic sclerosis as measured by the Short Form 36: relationship with clinical and biologic markers. Arthritis Rheum. 2004 Jun 15;51(3):475-81. doi: 10.1002/art.20389. PMID 15188336
- [Derived] Park EH, Strand V, Oh YJ, Song YW, Lee EB. Health-related quality of life in systemic sclerosis compared with other rheumatic diseases: a cross-sectional study. Arthritis Res Ther. 2019 Feb 15;21(1):61. doi: 10.1186/s13075-019-1842-x. PMID 30770765